CLINICAL TRIAL: NCT03945123
Title: Effect of Korea Red Ginseng on Non-alcoholic Fatty Liver Disease
Brief Title: Effects of Red Ginseng on Liver Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Ki Tae Suk, Proffesor, Chuncheon Sacred Heart Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIVER
Record Dates: First submitted 2019-05-03; First posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Liver Dysfunction
Keywords: ginseng; Liver
MeSH Terms: conditions — Liver Diseases | interventions — Asian ginseng

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ginseng trial (Experimental): compare experimental group to controlled group
  Interventions: Dietary Supplement: Red ginseng

INTERVENTIONS:
Dietary Supplement: Red ginseng — Red ginseng tablet 120g
  Other Names: Red ginseng tablet

SUMMARY:
Korea Red Ginseng (KRG) has effect on liver function

DETAILED DESCRIPTION:
Korea Red Ginseng (KRG) has been known as a natural product with anti-inflammatory effect in liver disease. Gut microbiota plays an important roles in the pathophysiology of nonalcoholic statohepatitis (NASH). We evaluated the effect of KRG on the pathophysiology of NASH

ELIGIBILITY:
Inclusion Criteria:

* AST or ALT level > 50 IU/L

Exclusion Criteria:

* Viral hepatitis
* Alcoholic hepatitis
* Autoimmune hepatitis
* Pancreatitis
* Hemochromatosis
* Wilson's disease
* Drug induced liver injury
* Cancer

Ages: 37 Years to 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Liver enzyme | 1year
  Decrease liver enzyme level

CONTACTS AND LOCATIONS:
Overall Officials: Ki Tae Suk, PhD.Md., Study Chair — Chuncheon Sacred Heart Hospital; Jun Seok, MD., Principal Investigator — Chuncheon Sacred Heart Hospital
Locations (1):
- ChuncheonSHH, Chuncheon, Gangwon-do, South Korea

IPD SHARING:
Plan to Share IPD: No
Not yet

REFERENCES:
- [Derived] Hong JT, Lee MJ, Yoon SJ, Shin SP, Bang CS, Baik GH, Kim DJ, Youn GS, Shin MJ, Ham YL, Suk KT, Kim BS. Effect of Korea red ginseng on nonalcoholic fatty liver disease: an association of gut microbiota with liver function. J Ginseng Res. 2021 Mar;45(2):316-324. doi: 10.1016/j.jgr.2020.07.004. Epub 2020 Jul 16. PMID 33841012